CLINICAL TRIAL: NCT06200454
Title: Predictive Value of Neuromuscular Ultrasound of Cranial Nerves in Guillain-Barré Syndrome
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, mohamed abdallah abdalraziq ahmed, resident doctor, Assiut University
Other Study IDs: U/S of cranial nerves in GBS
Record Dates: First submitted 2023-12-28; First posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2023-12

CONDITIONS: Guillain-Barre Syndrome
MeSH Terms: conditions — Guillain-Barre Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Guillain-Barré syndrome patients: neuromuscular ultrasound of cranial nerves
  Interventions: Device: neuromuscular ultrasound of cranial nerves
- normal participants: neuromuscular ultrasound of cranial nerves
  Interventions: Device: neuromuscular ultrasound of cranial nerves

INTERVENTIONS:
Device: neuromuscular ultrasound of cranial nerves — neuromuscular ultrasound of cranial nerves.

SUMMARY:
1. Sensitivity and specificity of cranial neuromuscular US to detect the prognosis of Guillain Barre Syndrome
2. Correlation of US values with motor, respiratory and autonomic complications of Guillain Barre Syndrome

DETAILED DESCRIPTION:
Guillain-Barré syndrome (GBS) is a dangerous and under certain circumstances life-threatening immune-mediated polyneuropathy of acute onset, often subsequent to respiratory or diarrheal illness. Patients usually present with distal onset of slight sensory symptoms such as numbness and tingling followed by ascending weakness of arms and legs, often involving cranial nerves Typical clinical findings are symmetric, flaccid paresis, reduced or absent deep tendon reflexes, and slight sensory symptoms only. Many variants of GBS such as pharyngeal-brachial or bulbar variants exist; the Miller-Fisher syndrome (MFS) with ataxia, areflexia, and oculomotor dysfunction; or the Elsberg syndrome with accentuated involvement of the autonomic nervous system. Diagnosis of GBS is normally based on typical clinical onset, laboratory findings, and electrophysiological studies.

In literature, Campylobacter jejuni infection is the most commonly identified precipitant of GBS. Cytomegalovirus, Epstein-Barr virus, human immunodeficiency virus (HIV), and Zika virus have also been reported with GBS [5]. A small percentage of patients develop GBS after other triggering events such as immunization, surgery, trauma, and bone-marrow transplantation.

Autonomic dysfunction (AD) in GBS predominantly occurs in the acute phase of the illness but can manifest in the recovery phase too. The exact mechanism remains unknown but probably involves dysfunction in the sympathetic and parasympathetic systems [8].

AD in GBS is observed in 70% of the cases [7]; features including tachycardia, bradycardia, facial flushing, hypertension alternating with hypotension, orthostatic hypotension, anhydrosis or diaphoresis, and urinary retention while gastrointestinal autonomic manifestation includes diarrhea or constipation [9]. Severe autonomic dysfunction is an important factor to recognize and treat accordingly as this is occasionally associated with a sudden death rate of 5-7% [10,11].

Guillain-Barré Syndrome (GBS) is often accompanied by respiratory failure that necessitates mechanical ventilation (MV).1 About 20-30% of cases require respiratory support.2-4 Major complications, including pulmonary infections, sepsis and pulmonary embolism, are reported in 60% of intubated patients with GBS.5, 6 The worldwide mortality rate for ventilated patients ranges from 15% to 30%, with survivors usually having poor outcomes.7 . Multiple clinical and biological parameters have been identified as risk factors for impending respiratory failure in GBS,9, 10 including cranial nerve involvement, disability grade on admission, rapidly progressive motor weakness, an absence of deep tendon reflexes, autonomic dysfunction, and features of nerve conduction block on electromyography.11-14

Facial nerve is commonly involved in GBS, occurring in at least half of patients. Other cranial nerves like bulbar nerves, abducent, oculomotor, optic, hypoglossal nerves are less often affected Ultrasound (US) is a reliable, effective, noninvasive, and well tolerated technique that allows multiple nerves to be examined in a relatively short period. Ultrasound (US) studies have demonstrated patchy enlargement of cranial nerves in Guillain-Barré syndrome (GBS). However, whether ultrasound yields useful information for early classification of GBS has not been established. We aimed to evaluate nerve ultrasound in patients with GBS in assuit university hospital. As confirmed in acquired immune-mediated neuropathies and inherited demyelinating neuropathies peripheral nerves can exhibit quantifiable enlargement in increased cross-sectional areas (CSA).

We follow up the patient to see improvement and accordingly we see the predictive value of neuromuscular ultrasound of cranial nerves in Guillain-Barré syndrome

ELIGIBILITY:
Inclusion Criteria:

* Patients fulfilling the diagnostic criteria of GBS within the first 2 weeks.
* Age: 18-65
* Both sexes

Exclusion Criteria:

* Past history of previous similar condition or history suggestive of CIDP.
* Any proved alternative diagnosis like hypo- or hyperkalemic paralysis, porphyria, or myositis.
* Other possible causes of peripheral neuropathy, diabetes, renal, and other metabolic disorders.
* History of Autonomic or cardiopulmonary dysfunction before the onset of symptoms.
* Patients who refused to participate or sign an informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Guillain-Barré syndrome (GBS) is a dangerous and under certain circumstances life-threatening immune-mediated polyneuropathy of acute onset, often subsequent to respiratory or diarrheal illness. Patients usually present with distal onset of slight sensory symptoms such as numbness and tingling followed by ascending weakness of arms and legs, often involving cranial nerves Typical clinical findings are symmetric, flaccid paresis, reduced or absent deep tendon reflexes, and slight sensory symptoms only. Many variants of GBS such as pharyngeal-brachial or bulbar variants exist; the Miller-Fisher syndrome (MFS) with ataxia, areflexia, and oculomotor dysfunction; or the Elsberg syndrome with accentuated involvement of the autonomic nervous system. Diagnosis of GBS is normally based on typical clinical onset, laboratory findings, and electrophysiological studies.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Estimated)
Dates: Start 2024-01-08 (Estimated); Primary Completion 2025-01-08 (Estimated); Study Completion 2025-06-08 (Estimated)

PRIMARY OUTCOMES:
Predictive value of neuromuscular ultrasound of cranial nerves in Guillain-Barré syndrome | baseline
  analysis of ultrasound results and follfow up of the cases to see if neuromuscular ultrasound of cranial nerves can predict the prognosis in Guillain-Barré syndrome

REFERENCES:
- [Background] Wilder-Smith EP. Swollen nerves slimming: Sequential nerve ultrasound in acute Guillain-Barre syndrome. Clin Neurophysiol. 2016 Feb;127(2):1013-1014. doi: 10.1016/j.clinph.2015.07.010. Epub 2015 Jul 17. No abstract available. PMID 26210255
- [Background] Abdelnaby R, Elsayed M, Mohamed KA, Dardeer KT, Sonbol YT, ELgenidy A, Barakat MH, NasrEldin YK, Maier A. Sonographic Reference Values of Vagus Nerve: A Systematic Review and Meta-analysis. J Clin Neurophysiol. 2022 Jan 1;39(1):59-71. doi: 10.1097/WNP.0000000000000856. PMID 34144573
- [Background] Guven SC, Bilgin E, Ozcakar L. Ultrasound imaging of the accessory nerve injury in a patient with thrombotic thrombocytopenic purpura and polyneuropathy. Am J Phys Med Rehabil. 2014 Oct;93(10):928. doi: 10.1097/PHM.0000000000000130. No abstract available. PMID 24919085
- [Background] Curcean AD, Rusu GM, Dudea SM. Ultrasound appearance of peripheral nerves in the neck: vagus, hypoglossal and greater auricular. Med Pharm Rep. 2020 Jan;93(1):39-46. doi: 10.15386/mpr-1273. Epub 2020 Jan 31. PMID 32133445